CLINICAL TRIAL: NCT02854033
Title: Alzheimer's Disease Neuroimaging Initiative 3 (ADNI3)
Acronym: ADNI3
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Northern California Institute of Research and Education (Other); National Institute on Aging (NIA) (NIH); Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Principal Investigator, Paul S. Aisen, Director, Alzheimer's Therapeutic Research Institute, University of Southern California
Other Study IDs: ATRI-001; U01AG024904 (NIH)
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment (MCI); Alzheimer's Disease (AD)
Keywords: amyloid; plaques; neuroimaging; biomarkers; cognition disorder; early detection; pre-dementia; dementia; Alzheimer's disease; tau
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Plaque, Amyloid; Cognition Disorders; Dementia; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cognitively Normal (CN): 135-500 newly enrolled participants with no apparent memory problems, and 295-300 cognitively normal participants followed from the ADNI2 study.
  Currently recruiting non-Caucasian participants only for the normal cognition group.
- Mild Cognitive Impairment (MCI): 150 - 515 newly enrolled participants with mild cognitive impairment (MCI), and 275-320 MCI participants followed from the ADNI2 study.
- Mild Alzheimer's Disease (AD) dementia: 85 - 185 newly enrolled participants with mild Alzheimer's disease (AD) dementia, and 130 - 150 mild AD participants followed from the ADNI2 study.

SUMMARY:
Since its launch in 2004, the overarching aim of the Alzheimer's Disease Neuroimaging Initiative (ADNI) has been realized in informing the design of therapeutic trials in AD. ADNI3 continues the previously funded ADNI-1, ADNI-GO, and ADNI-2 studies that have been combined public/private collaborations between academia and industry to determine the relationships between the clinical, cognitive, imaging, genetic and biochemical biomarker characteristics of the entire spectrum of Alzheimer's disease (AD). The overall goal of the study is to continue to discover, optimize, standardize, and validate clinical trial measures and biomarkers used in AD research.

DETAILED DESCRIPTION:
The overall goal of ADNI3 is to determine the relationships among the clinical, cognitive, imaging, genetic and biochemical biomarker characteristics of the entire spectrum of Alzheimer's disease (AD), as the pathology evolves from normal aging through very mild symptoms, to mild cognitive impairment (MCI), to dementia. ADNI3 continues the previously funded AD Neuroimaging Initiative (ADNI1, ADNI-GO, and ADNI-2), and remains a public/private collaboration between academia and industry to study biomarkers of AD. ADNI will continue to inform the neuroscience of AD, identify diagnostic and prognostic markers, identify outcome measures that can be used in clinical trials, and help develop the most effective clinical trial scenarios.

This is multi-center, a non-randomized, natural history, non-treatment study. 1,070-2,000 total participants will be enrolled across three cohorts: cognitively normal* (CN), mild cognitive impairment (MCI) and mild Alzheimer's Disease (AD) dementia. Participants between the ages of 55-90 (inclusive) will be enrolled at 59 sites in the United States and Canada. Approximately, 700 - 800 will be rollover participants from previous ADNI studies, and 370 - 1200 will be newly enrolled. Clinical/cognitive, imaging, biomarker, and genetic characteristics will be assessed across the three cohorts.

Participants will undergo longitudinal clinical and cognitive assessments, computerized cognitive batteries, biomarker and genetic tests, PET (FDG, amyloid and tau) and MRI scans and cerebral spinal fluid (CSF) collection for up to 5 years.

*currently recruiting non-Caucasian participants only for the cognitively normal cohort.

ELIGIBILITY:
Inclusion Criteria (all CN participants):

1. Participant with or without subjective memory complaints, verified by a study partner, beyond what one would expect for age
2. Normal memory function documented by scoring above education adjusted cutoffs on the Logical Memory II subscale (Delayed Paragraph Recall, Paragraph A only) from the Wechsler Memory Scale -Revised (the maximum score is 25):

   1. 9 for 16 or more years of education
   2. 5 for 8-15 years of education
   3. 3 for 0-7 years of education
3. Mini-Mental State Exam score between 24 and 30 inclusive (Exceptions may be made for participants with less than 8 years of education at the discretion of the Project Director)
4. Clinical Dementia Rating = 0. Memory Box score must be 0
5. Cognitively normal, based on an absence of significant impairment in cognitive functions or activities of daily living
6. Stability of Permitted Medications for at least 4 weeks:

   1. Stable doses of antidepressants lacking significant anticholinergic side effects (if they are currently adequately treated for depressive symptoms and do not have a history of major depression within the past 1 years)
   2. Estrogen replacement therapy is permissible
   3. Gingko biloba is permissible, but discouraged
   4. Washout from psychoactive medication (e.g., excluded antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.) for at least 4 weeks prior to screening.

Inclusion Criteria (all MCI participants):

1. Participant must express a subjective memory concern as reported by participant, or recalled by study partner or clinician.
2. Abnormal memory function documented by scoring below education adjusted cutoffs on the Logical Memory II subscale (Delayed Paragraph Recall, Paragraph A only) from the Wechsler Memory Scale -Revised (the maximum score is 25):

   a. < 11 for 16 or more years of education b. ≤ 9 for 8-15 years of education c. ≤ 6 for 0-7 years of education
3. Mini-Mental State Exam score between 24 and 30 inclusive (Exceptions may be made for participants with less than 8 years of education at the discretion of the Project Director)
4. Clinical Dementia Rating = 0.5. Memory Box score must be at least 0.5
5. General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's disease cannot be made by the site physician at the time of the Screening Visit
6. Stability of Permitted Medications for at least 4 weeks:

   1. Stable doses of antidepressants lacking significant anticholinergic side effects (if they are currently adequately treated for depressive symptoms and do not have a history of major depression within the past 1 years)
   2. Cholinesterase inhibitors and memantine are allowable if stable for 12 weeks prior to Screening Visit
   3. Estrogen replacement therapy is permissible
   4. Gingko biloba is permissible, but discouraged
   5. Washout from psychoactive medication (e.g., excluded antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.) for at least 4 weeks prior to screening.

Inclusion Criteria (all AD participants):

1. Participant must express a subjective memory concern as reported by participant, or recalled by study partner or clinician.n.
2. Abnormal memory function documented by scoring below education adjusted cutoffs on the Logical Memory II subscale (Delayed Paragraph Recall, Paragraph A only) from the Wechsler Memory Scale -Revised (the maximum score is 25):

   1. ≤ 8 for 16 or more years of education
   2. ≤ 4 for 8-15 years of education
   3. ≤ 2 for 0-7 years of education
3. Mini-Mental State Exam score between 20 and 26 inclusive (Exceptions may be made for participants with less than 8 years of education at the discretion of the Project Director)
4. Clinical Dementia Rating = 0.5 or 1.0
5. NINCDS (National Institute of Neurological and Communicative Disorders and Stroke) -ADRDA (Alzheimer's Disease and Related Disorders Association) criteria for probable AD
6. Stability of Permitted Medications for at least 4 weeks:

   1. Stable doses of antidepressants lacking significant anticholinergic side effects (if they are currently adequately treated for depressive symptoms and do not have a history of major depression within the past 1 years)
   2. Cholinesterase inhibitors and memantine are allowable if stable for 12 weeks prior to Screening Visit
   3. Estrogen replacement therapy is permissible
   4. Gingko biloba is permissible, but discouraged
   5. Washout from psychoactive medication (e.g., excluded antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.) for at least 4 weeks prior to screening.

Inclusion Criteria Specific to Newly Enrolled Participants

1. Geriatric Depression Scale score less than 6.
2. Age between 55-90 years (inclusive).
3. Study partner who has frequent contact with the participant (i.e., minimum average of 10 hours per week) and is available to accompany the participant to all clinic visits for the duration of the protocol.
4. Visual and auditory acuity adequate for neuropsychological testing.
5. Good general health with no diseases expected to interfere with the study.
6. Participant is not pregnant, lactating, or of childbearing potential (i.e. women must be two years post-menopausal or surgically sterile).
7. Willing and able to participate in a longitudinal imaging study.
8. Modified Hachinski Ischemic Score less than or equal to 4.
9. Completed six grades of education or has a good work history (sufficient to exclude mental retardation).
10. Must speak English or Spanish fluently.
11. Willing to undergo repeated MRIs (3Tesla) and at least two PET scans
12. Agrees to collection of blood for genomic analysis (including GWAS (genome-wide association study) sequencing and other analysis), APOE (Apolipoprotein E) testing and biospecimen banking.
13. Agrees to collection of blood for biomarker testing.
14. Agrees to at least one lumbar puncture for the collection of CSF.
15. Agrees to share genomic data and biomarker samples. Inclusion Criteria Specific to Rollover Participants"

The following additional inclusion criteria apply to all diagnostic categories for rollover participants only:

1. Must have been enrolled and followed in ADNI-1, ADNI-GO, or ADNI-2 for at least one year.
2. Willing and able to continue to participate in an ongoing longitudinal study. A reduced battery of tests is allowable if the participant is not able/willing to complete the full battery.

Exclusion Criteria (all CN participants):

1. Any significant neurologic disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities

Exclusion Criteria (all MCI participants):

1. Any significant neurologic disease other than suspected incipient Alzheimer's disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.

Exclusion Criteria (all AD participants):

1. Any significant neurologic disease other than Alzheimer's disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.

Exclusion Criteria (all participants):

The following additional exclusion criteria apply to all diagnostic categories:

1. Screening/Baseline MRI brain scan with evidence of infection, infarction, or other focal lesions or multiple lacunes or lacunes in a critical memory structure
2. Subjects that have any contraindications for MRI studies, including the presence of cardiac pacemakers, or metal fragments or foreign objects in the eyes, skin or body.
3. Major depression, bipolar disorder as described in DSM-IV within the past 1 year. Psychotic features, agitation or behavioral problems within the last 3 months that could lead to difficulty complying with the protocol.
4. Currently treated with medication for obsessive-compulsive disorder or attention deficit disorder.
5. History of schizophrenia (DSM IV criteria).
6. History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
7. Any significant systemic illness or unstable medical condition, which could lead to difficulty complying with the protocol.
8. Clinically significant abnormalities in B12 or thyroid function tests (TFTs) that might interfere with the study. A low B12 is exclusionary, unless follow-up labs (homocysteine (HC) and methylmalonic acid (MMA)) indicate that it is not physiologically significant.
9. Residence in a skilled nursing facility.
10. Current use of specific psychoactive medications (e.g., certain antidepressants, neuroleptics, chronic anxiolytics or sedative hypnotics). Current use of warfarin or other anticoagulants such as dabigatran, rivaroxaban and apixaban (exclusionary for lumbar puncture).
11. Current use of any other exclusionary medications
12. Investigational agents are prohibited one month prior to entry and for the duration of the trial.
13. Participation in clinical studies involving neuropsychological measures being collected more than one time per year.

Exclusion Criteria Specific to AV-1451 PET:

The following criteria are exclusionary only for the AV-1451 scanning portion of the study:

1. History of risk factors for torsades de pointes (a cardiac dysrhythmia associated with sudden death) or taking medications known to prolong the QT interval. A list of restricted medications will be provided.
2. Have an ECG obtained prior to the AV-1451 PET scan that in the opinion of the investigator is clinically significant with regard to the subject's participation in the study. Bazett's corrected QT (QTcB) interval must be evaluated and must not exceed 458 msec in males, or 474 msec in females.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cognitively normal (CN), mild cognitive impairment (MCI), and mild AD dementia participants.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-10; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of change in cognition as measured by the Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog13) | 5 years
  The ADAS-Cog is an in-person examiner-administered, structured scale that evaluates memory (word recall, word recognition), reasoning (following commands), language (naming, comprehension), orientation, ideational praxis (placing letter in envelope) and constructional praxis (copying geometric designs). Ratings of spoken language, language comprehension, word finding difficulty, and ability to remember test instructions are also obtained.
Rate of change in cognition as measured by the Logical Memory Test I and II | 5 years
Rate of change in cognition as measured by the Mini-Mental State Examinations (MMSE) | 5 years
  The MMSE scale evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two overlapping pentagons.

SECONDARY OUTCOMES:
Rate of change in cognition as measured by the Cogstate Brief Battery (CBB) | 5 years
  The Cogstate Brief battery (CBB) is a brief (10-15 minute) computerized cognitive battery developed by Cogstate (Cogstate Ltd. New Haven, CT, USA) that measures attention, speed of information processing, working memory and learning.
Rate of change in cognition as measured by the American National Adult Reading Test (ANART) | 5 years
  The ANART estimates premorbid verbal intelligence (VIQ) in patients with dementia.
Rate of change in cognition as measured by the Montreal Cognitive Assessment (MoCA) | 5 years
  The Montreal Cognitive Assessment test (MoCA) is a cognitive assessment designed to detect participants at the MCI stage of cognitive dysfunction.
Rate of change in cognition as measured by the Rey Auditory Verbal Learning Test | 5 years
  The AVLT is a list-learning task, which assesses multiple cognitive parameters associated with learning and memory.
Rate of change in cognition as measured by the Trail Making Test: A and B | 5 years
Change in tau deposition as measured by 18F-AV-1451 | 5 years
Change in amyloid deposition as measured by Florbetapir | 5 years
Change in amyloid deposition as measured by Florbetaben | 5 years
Rate of conversion to MCI or dementia due to AD | 5 years
Rates of change of glucose metabolism (FDG-PET) | 5 years
Change in Cerebral Spinal Fluid (CSF) Tau Biomarkers | 5 years
Change in brain structure using magnetic resonance imaging (MRI) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Weiner, MD, Study Director — University of California, San Francisco; Paul Aisen, MD, Principal Investigator — USC Alzheimer's Therapeutic Research Institute (ATRI); Ronald Peterson, MD, PHD, Principal Investigator — Mayo Clinic
Locations (59):
- United States (54):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California, Irvine, Irvine, California
  - University of California, San Diego, La Jolla, California
  - Long Beach VA Neuropsychiatric Research Program, Long Beach, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - VA Palo Alto HSC / Stanford School of Medicine, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - University of California, Davis, Walnut Creek, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Wien Center for Clinical Research, Miami Beach, Florida
  - University of South Florida - Health Byrd Alzheimer Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Fairway, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Albany Medical College, Albany, New York
  - Dent Neurologic Institute, Buffalo, New York
  - New York University Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - Nathan Kline Institute for Psychiatric Research, Orangeburg, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Beachwood, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital Memory and Aging Program, Providence, Rhode Island
  - Ralph H. Johnson VA Health Care System, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, Southwestern MC at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Canada (5):
  - University of British Columbia, Clinic for AD & Related, Vancouver, British Columbia
  - Parkwood Institute, London, Ontario
  - St. Joseph's Health Center - Cognitive Neurology, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital Memory Clinic, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Miller AA, Sharp ES, Wang S, Zhao Y, Mecca AP, van Dyck CH, O'Dell RS; Alzheimer's Disease Neuroimaging Initiative (ADNI). Self-reported hearing loss is associated with faster cognitive and functional decline but not diagnostic conversion in the ADNI cohort. Alzheimers Dement. 2024 Nov;20(11):7847-7858. doi: 10.1002/alz.14252. Epub 2024 Sep 26. PMID 39324520
- [Derived] Howe MD, Caruso MR, Manoochehri M, Kunicki ZJ, Emrani S, Rudolph JL, Huey ED, Salloway SP, Oh H; Alzheimer's Disease Neuroimaging Initiative. Utility of cerebrovascular imaging biomarkers to detect cerebral amyloidosis. Alzheimers Dement. 2024 Oct;20(10):7220-7231. doi: 10.1002/alz.14207. Epub 2024 Sep 1. PMID 39219209
- [Derived] Howe MD, Caruso MR, Manoochehri M, Kunicki ZJ, Emrani S, Rudolph JL, Huey ED, Salloway SP, Oh H; Alzheimer's Disease Neuroimaging Initiative. Utility of cerebrovascular imaging biomarkers to detect cerebral amyloidosis. medRxiv [Preprint]. 2024 May 28:2024.05.28.24308056. doi: 10.1101/2024.05.28.24308056. PMID 38853879
- [Derived] Rauchmann BS, Schneider-Axmann T, Perneczky R; Alzheimer's Disease Neuroimaging Initiative (ADNI). Associations of longitudinal plasma p-tau181 and NfL with tau-PET, Abeta-PET and cognition. J Neurol Neurosurg Psychiatry. 2021 Dec;92(12):1289-1295. doi: 10.1136/jnnp-2020-325537. Epub 2021 Jun 29. PMID 34187867
- [Derived] Bullich S, Roe-Vellve N, Marquie M, Landau SM, Barthel H, Villemagne VL, Sanabria A, Tartari JP, Sotolongo-Grau O, Dore V, Koglin N, Muller A, Perrotin A, Jovalekic A, De Santi S, Tarraga L, Stephens AW, Rowe CC, Sabri O, Seibyl JP, Boada M. Early detection of amyloid load using 18F-florbetaben PET. Alzheimers Res Ther. 2021 Mar 27;13(1):67. doi: 10.1186/s13195-021-00807-6. PMID 33773598
- See also: Alzheimer's Disease Neuroimaging Initiative — http://adni-info.org
- See also: Laboratory of Neuro Imaging (LONI) — http://adni.loni.usc.edu/
- See also: Alzheimer's Therapeutic Research Institute — http://atri.usc.edu/studies/
- See also: List of Alzheimer's Disease Neuroimaging Initiative Publications — http://adni.loni.usc.edu/news-publications/publications/
- See also: Brain Health Registry (BHR) — http://www.brainhealthregistry.org/